CLINICAL TRIAL: NCT00039234
Title: A Phase III, Multi-Center Controlled Trial With Stratified Randomization Comparing The Efficacy Of Interleukin-2 (IL-2) Plus Histamine Dihydrochloride (HDC) Versus IL-2 Alone To Increase The Duration Of Survival In Patients With AJCC Stage IV Malignant Melanoma With Hepatic Metastasis
Brief Title: Interleukin-2 With or Without Histamine Dihydrochloride in Treating Patients With Stage IV Melanoma Metastatic to the Liver
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maxim Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069365; MAXIM-MP-8899-0104; UCLA-0111056; NCI-G02-2070; MSKCC-03057
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2003-12

CONDITIONS: Melanoma (Skin); Metastatic Cancer
Keywords: stage IV melanoma; recurrent melanoma; liver metastases
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — aldesleukin; Histamine

INTERVENTIONS:
Biological: aldesleukin
Drug: histamine dihydrochloride

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Histamine dihydrochloride may help interleukin-2 kill more tumor cells by making tumor cells more sensitive to the drug. It is not yet known if interleukin-2 is more effective with or without histamine dihydrochloride in treating stage IV melanoma that is metastatic to the liver.

PURPOSE: Randomized phase III trial to compare the effectiveness of interleukin-2 with or without histamine dihydrochloride in treating patients who have stage IV melanoma that is metastatic to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the duration of survival in patients with stage IV melanoma with hepatic metastasis treated with interleukin-2 with or without histamine dihydrochloride.
* Compare the progression-free survival, response rate, response rate of hepatic tumors, and lack of disease progression in patients treated with these regimens.
* Determine the safety of these regimens, in terms of frequency, severity, and causal relationship of adverse events, in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center location (North America vs Europe), lactate dehydrogenase (less than ULN vs ULN or greater), and metastatic sites (liver only vs liver and other sites). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive interleukin-2 (IL-2) subcutaneously (SC) twice daily on days 1 and 2 of weeks 1 and 3 and days 1-5 of weeks 2 and 4. Patients also receive histamine dihydrochloride SC over 10-30 minutes on days 1-5 of weeks 1-4.
* Arm II: Patients receive IL-2 as in arm I. In both arms, treatment repeats every 6 weeks for at least 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 3 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 224 patients (112 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma

  * Must have radiological evidence of lesions in liver (target or non-target)
* At least 1 measurable lesion outside previously irradiated field

  * At least 20 mm by contrast-enhanced CT scan, MRI, medical photography, or physical exam OR at least 10 mm by spiral CT scan
* No prior or concurrent clinical and/or objective evidence of brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 9.5 g/dL
* WBC at least 3,000/mm^3
* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT no greater than 4 times ULN
* Alkaline phosphatase no greater than 4 times ULN
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 1.7 mg/dL
* Calcium no greater than 11.5 mg/dL

Cardiovascular:

* No abnormal thallium stress test
* No acute myocardial infarction within the past year
* No New York Heart Association class III or IV heart disease

Pulmonary:

* No asthma requiring active treatment within the past 5 years
* Oxygen saturation by pulse oximeter at least 90% unless FEV_1 is greater than 2 L or at least 75% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Concurrent medically-controlled (except with glyburide) or diet-controlled diabetes is allowed
* Concurrent medically-controlled thyroid dysfunction is allowed
* No other active malignancy within the past 5 years except carcinoma in situ of the cervix or localized squamous cell or basal cell skin cancer
* No serious non-malignant medical conditions, including psychiatric disability, that would preclude study compliance
* No active autoimmune disease (e.g., lupus, inflammatory bowel disease, or psoriasis)
* No active peptic and/or esophageal ulcer disease
* No hypersensitivity to histamine products or urticaria
* No active IV drug abuse

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy with high-dose IV interleukin-2 (IL-2)
* No prior combination immunotherapy with chemotherapy
* At least 1 year since prior low-dose adjuvant IL-2 as part of vaccine therapy or as therapy for stage II or III melanoma

Chemotherapy:

* See Biologic therapy

Endocrine therapy:

* No chronic systemic glucocorticoid steroids

  * Asthma inhalers, topical creams, or intra-articular injections allowed
* Hormonal therapy for non-melanoma-related conditions allowed

Radiotherapy:

* See Disease Characteristics
* Concurrent radiotherapy as palliative therapy for isolated non-target lesions (e.g., bone lesions) allowed

Surgery:

* Not specified

Other:

* At least 4 weeks since prior therapy directed at malignancy
* At least 4 weeks since prior investigational medications or therapies
* At least 2 weeks since prior parenteral antioxidants and/or vitamins
* At least 2 weeks since prior antibiotics for active illness
* At least 2 weeks since prior H2 antagonists, beta-blockers, antihypertensives, antimalarials, antitrypanosomals, neuromuscular-blocking agents, tricyclic antidepressants, or alprazolam
* At least 24 hours since prior antihistamines
* No prior enrollment in any Maxim Pharmaceuticals investigational trials
* No concurrent anticonvulsant therapy for seizure disorder
* No other concurrent investigational drug
* No concurrent H2 antagonists, tricyclic antidepressants, alprazolam, beta- blockers, antihypertensives, antitrypanosomals, antimalarials, or monoamine oxidase inhibitors
* No concurrent inhibitors of diamine oxidase, monoamine oxidase, or histamine N-methyltransferase
* No concurrent antihistamines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Study Chair — Jonsson Comprehensive Cancer Center
Locations (19):
- United States (11):
  - John Wayne Cancer Institute at Saint John's Health Center, Santa Monica, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Moffitt Clinic at Tampa General Hospital, Tampa, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Melanoma Center of St. Louis, Missouri Baptist Medical Center, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Comprehensive Cancer Center at Our Lady of Mercy Medical Center, The Bronx, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- Germany (5):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Universitatsklinik - Saarland, Homburg/Saar
  - Kiel Universitatshautklinik, Kiel
  - Klinische Kooperationseinheit fur Dermatoonkologie (DFKZ), Mannheim
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich
- Royal Marsden Hospital - Sutton, London, England, United Kingdom